CLINICAL TRIAL: NCT03979729
Title: Breast Cancer Screening Among Medically Underserved Women in New Mexico: Comparing Outcomes and LOwering Recall Rates With Digital Breast Tomosynthesis (3D Mammography) VErsus Full-field Digital (2D) Mammography. The LOVE New Mexico Study
Brief Title: Breast Cancer Screening for Underserved Women: Comparing Outcomes and Lowering Recall Rates With 3D- vs. 2D-mammography
Status: Completed | Type: Observational
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: INST UNM 1525
Record Dates: First submitted 2019-05-13; First posted 2019-06-07 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 3D + 2D-Mammogram Recipients (Patient Group A): Women presenting for mammographic screening who selected 3D + 2D- mammogram. These women will undergo in-person or telephone interviews.
  Interventions: Other: Routine Screening Mammogram (3D + 2D)
- 2D-Mammogram Recipients (Patient Group B): Women presenting for mammographic screening who selected 2D- mammogram alone (declined 3D + 2D- mammogram). These women will undergo in-person or telephone interviews.
  Interventions: Other: Routine Screening Mammogram (2D)
- Women Who Have Never Received a Mammogram (Patient Group C): Women who have never undergone recommended mammographic screening. These women will participate in a onetime facilitated focus group.
  Interventions: Other: No Screening Mammogram
- Providers: Primary care providers (physicians, physicians assistants, and advanced nurse practitioners) working in clinics providing primary care for underserved patient populations in New Mexico, including primary care providers at a RIOSNET-affiliated and UNM-affiliated clinics

INTERVENTIONS:
Other: Routine Screening Mammogram (3D + 2D) — Subjects that have undergone a routine screening mammogram (3D + 2D) will be interviewed by a member of the research team who will ask a few questions to better understand how the subject made this decision and what things may have influenced her decision between different types of mammograms.
  Groups: 3D + 2D-Mammogram Recipients (Patient Group A)
Other: Routine Screening Mammogram (2D) — Subjects that have undergone a routine screening mammogram (2D) will be interviewed by a member of the research team who will ask a few questions to better understand how the subject made this decision and what things may have influenced her decision between different types of mammograms.
  Groups: 2D-Mammogram Recipients (Patient Group B)
Other: No Screening Mammogram — Subjects will participate in a one-time facilitated focus group.
  Groups: Women Who Have Never Received a Mammogram (Patient Group C)

SUMMARY:
Three-dimensional (3D) + two-dimensional (2D)- mammography may have particular value for minority, rural, and underserved women in New Mexico by decreasing recall rates and improving diagnostic sensitivity, thus alleviating some of the unique burdens associated with breast cancer screening in the multi-ethnic and underserved New Mexico patient population. Primary objective: To compare recall rates using 3D + 2D- vs. 2D- mammogram in New Mexico women undergoing screening mammogram between 2013 and 2016. Secondary objectives: Evaluate knowledge, attitudes, perceived barriers, intentions, decisional influences, and other psychosocial/cultural factors influencing breast cancer screening among medically underserved patients and assess what impact 3D + 2D-mammography might have on those perceptions; Determine primary care providers' knowledge, attitudes, beliefs, and preferences regarding 3D + 2D- vs. 2D- mammography; evaluate breast cancer detection rate and biopsy positive predictive value for screening mammograms using 3D + 2D- vs. 2D using PENRAD data; evaluate screening outcome, compliance with recall recommendations, breast cancer detection rate, positive predictive value, and demographics of interest in New Mexico women undergoing screening and offered 3-D mammography (retrospective chart review).

DETAILED DESCRIPTION:
This project will have both a prospective and retrospective component.

Retrospective component:

Primary Objective: To compare recall rates using 3D + 2D- vs. 2D mammogram in New Mexico women undergoing screening mammograms between 2013 and 2016. Data abstraction from the PENRAD database will be completed by staff in the Department of Radiology. Data abstraction for the chart review of the subgroup of State-funded patients will be conducted with HIPAA-compliant practices from the University of New Mexico Hospital (UNMH) electronic medical record. Data analysis will be performed by study investigators.

Prospective component:

Secondary Objective 1: To evaluate knowledge, attitudes, perceived barriers, intentions, and decisional influences (conflict, regret, satisfaction), and other psychosocial/cultural factors influencing breast cancer screening (including concerns over recall vs. radiation exposure) among medically underserved patients and to assess what impact 3D + 2D-mammography (with a potentially lower recall rate but higher radiation exposure) might have on those perceptions. Patients in Groups A and B will undergo 1:1 interviews. Patients in Group C will participate in a one-time focus group (6-8 women per group).

Secondary Objective 2: To determine primary care providers' knowledge, attitudes, beliefs, and preferences regarding 3D + 2D vs. 2D- mammography. Providers will undergo interviews.

Secondary Objective 3A: To evaluate breast cancer detection rate and biopsy positive predictive value in New Mexico women undergoing screening mammogram using 3D + 2D- vs. 2D- mammogram using PENRAD data collected from the group as a whole. This objective will be met via database query alone. No individual mammographic images will be evaluated.

Secondary Objective 3B: To evaluate screening outcome, compliance with recall recommendations, breast cancer detection rate, positive predictive value, and demographics of interest in New Mexico women undergoing screening and offered 3-D mammography using retrospective chart review. Demographic variables will include age, self-reported ethnicity, city of residence, and health insurance type. This objective will be met via database query alone. No individual mammographic images will be evaluated.

ELIGIBILITY:
Inclusion Criteria for Retrospective Component (Primary Objective):

* Screening mammographic examinations performed in women over age 40 undergoing 3D +2D- or 2D-screening mammogram through the University of New Mexico's Department of Radiology at the University of New Mexico Hospital (UNMH) and Sandoval Regional Medical Center (SRMC) between 2013 and 2016

Inclusion Criteria for Prospective Component (Secondary Objective #1) (Patient Groups A and B)

* Women over age 40 undergoing screening mammogram through the University of New Mexico's Department of Radiology as recommended and ordered by their primary care provider
* Must have the ability to understand a consent form
* Enrolled or eligible for the Department of Health / State of New Mexico Breast and Cervical Cancer Screening Program or Medicaid
* Must have been offered a choice of either 3D + 2D-mammography or 2D-mammography as screening for breast cancer and underwent the selected screening prior to consent
* Pregnant women may participate in this study

Exclusion Criteria for Prospective Component (Secondary Objective #1) (Patient Groups A and B):

* Cognitively impaired adult women are excluded from participation
* Adult women not able to consent for themselves are excluded from participation
* Prisoners may not participate in this study

Inclusion Criteria for Prospective Component (Secondary Objective #1) (Patient Group C):

* Women over age 40 recommended for mammographic screening for breast cancer by a primary care provider, but have never completed a screening mammogram
* Must have the ability to understand a consent form
* Enrolled or eligible for the Department of Health / State of New Mexico Breast and Cervical Cancer Screening Program or for Medicaid
* Pregnant women may participate in this study

Exclusion Criteria for Prospective Component (Secondary Objective #1) (Patient Group C):

* Cognitively impaired adult women are excluded from participation
* Adult women not able to consent for themselves are excluded from participation
* Prisoners may not participate in this study

Inclusion Criteria for Providers (Secondary Objective #2):

* Primary care providers (physicians, physicians assistants, and advanced nurse practitioners) working in clinics providing primary care for underserved patient populations in New Mexico, including primary care providers at a RIOSNET-affiliated and UNM-affiliated clinics

Exclusion Criteria for Providers (Secondary Objective #2):

* Any primary care provider who does not order screening mammography for eligible participants or is under Medicaid violation review

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Retrospective and prospective portions of study (patients): Women over age 40 recommended for mammographic screening for breast cancer by a primary care provider, who are enrolled or eligible for the Department of Health / State of New Mexico Breast and Cervical Cancer Screening Program or Medicaid.
  Prospective portion (providers): Primary care providers (physicians, physicians assistants, and advanced nurse practitioners) working in clinics providing primary care for underserved patient populations in New Mexico, including primary care providers at a RIOSNET-affiliated and UNM-affiliated clinics.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2016-09-22 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
Recall rates using 3D + 2D- vs. 2D-mammogram in New Mexico women undergoing screening mammograms (Retrospective analysis) | 5 years
  Compare the recall rates of New Mexico (NM) women over age 40 who underwent 3D + 2D screening mammograms vs. recall rates for women who underwent 2D- screening mammograms between 2013 and 2016 through the University of New Mexico's Department of Radiology at the University of New Mexico Hospital (UNMH) and Sandoval Regional Medical Center (SRMC). The "recall rate" is defined as the percentage (number of patients recalled per 100 patients who had mammograms) of New Mexico women undergoing screening mammogram between 2013 and 2016 recalled for additional diagnostic imaging when screening mammogram was performed with digital breast tomosynthesis (3D + 2D-mammography) or 2- dimensional full-field digital mammography alone. The University of New Mexico's Department of Radiology PENRAD database will queried anonymously for this data.

SECONDARY OUTCOMES:
What psychosocial and cultural factors influence breast cancer screening among medically underserved patients, identified through interviews and questionnaires | 5 years
  Use interviews to create qualitative (descriptive) assessments of the knowledge, attitudes, perceived barriers, intentions, and decisional influences (conflict, regret, satisfaction), and other psychosocial/cultural factors influencing breast cancer screening (including concerns over recall vs. radiation exposure) among medically underserved patients enrolled in or eligible for the Department of Health / State of New Mexico Breast and Cervical Cancer Screening Program or Medicaid and to assess what impact 3D + 2D-mammography (with a potentially lower recall rate but higher radiation exposure) might have on those perceptions.
What are primary care providers' knowledge, attitudes, beliefs, and preferences regarding 3D + 2D- vs. 2D-mammography, identified through interviews and questionnaires | 5 years
  Use interviews to create qualitative (descriptive) assessments of care providers' knowledge, attitudes, beliefs, and preferences regarding 3D + 2D- vs. 2D-mammography.
Breast cancer detection rate for 3D + 2D- vs. 2D-mammograms | 5 years
  Evaluate breast cancer detection rate (per 100 patients, percentage) in New Mexico women undergoing screening mammograms using 3D + 2D- vs. 2D-mammogram using PENRAD (mammography tracking software) data collected from the group as a whole.
Breast cancer biopsy positive predictive value for 3D + 2D- vs. 2D-mammograms | 5 years
  Evaluate breast cancer biopsy positive predictive value (per 1000 patients) in New Mexico women undergoing screening mammograms using 3D + 2D- vs. 2D-mammogram using PENRAD (mammography tracking software) data collected from the group as a whole.
Screening outcome of women undergoing 3-D mammography | 5 years
  Evaluate screening outcome in New Mexico women undergoing screening and offered 3-D mammography based on eligibility requirements for NM House Bill 2, using retrospective chart review.
Compliance with recall recommendations of women undergoing 3-D mammography | 5 years
  Evaluate compliance with recall recommendations in New Mexico women undergoing screening and offered 3-D mammography based on eligibility requirements for NM House Bill 2, using retrospective chart review.
Breast cancer detection rate in women undergoing 3-D mammography | 5 years
  Evaluate breast cancer detection rate (per 100 patients) of New Mexico women undergoing screening and offered 3-D mammography based on eligibility requirements for NM House Bill 2, using retrospective chart review.
Positive predictive value of women undergoing 3-D mammography | 5 years
  Evaluate positive predictive value (per 1000 patients) in New Mexico women undergoing screening and offered 3-D mammography based on eligibility requirements for NM House Bill 2, using retrospective chart review.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Fine, MD, Principal Investigator — University of New Mexico Comprehensive Cancer Center
Locations (1):
- University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Manda-Mapalo MT, Fine SG, Safadi S, Lee JH, Du R, Sussman AL, Mishra S, Selwyn RG, Saline JL, Hine WL, Brown-Glaberman UA. Breast Cancer Screening Among Medically Underserved Women in New Mexico: Potential for Lower Recall Rates with Digital Breast Tomosynthesis. J Womens Health (Larchmt). 2020 Dec;29(12):1596-1601. doi: 10.1089/jwh.2020.8402. Epub 2020 Sep 29. PMID 32991242